CLINICAL TRIAL: NCT00309816
Title: Measurement of the Effect of Sildenafil Citrate (Viagra) on the Hemodynamics of Exercise Tolerance in Advanced Congestive Heart Failure.
Brief Title: Study of Sildenafil in Patient With Heart Failure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001-p-001039
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Congestive Heart Failure
Keywords: Exercise stress test
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
The purpose of this study is to determine if sildenafil (Viagra) improves exercise tolerance.

DETAILED DESCRIPTION:
Patients will undergo an exercise stress test. One dose of Sildenafil will then be given, followed by a one hour rest period. A repeat exercise stress test will then be repeated.

ELIGIBILITY:
Inclusion Criteria:

Age 18 - 75 Ejection fraction <35% Heart failure limited by fatigue and shortness of breath -

Exclusion Criteria:

Inability to exercise. Patients with shortness of breath while resting. Patient requiring intravenous medication. Patients taking the following medications: nitroglycerine pill/patch/paste, isordil and Imdur

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Patients will have exercise capacity measured by an exercise stress test before and after one dose of sildenafil.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Semigran, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States